CLINICAL TRIAL: NCT03211000
Title: Study of the Molecular Mechanisms Associated With the Formation of Human Aortic Aneurysm: a Focus on Autophagy, Oxidative Stress and Hippo Signaling
Brief Title: Autophagy, Oxidative Stress and Hippo Signaling in Human Aortic Aneurysm
Status: Completed | Type: Observational
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Maurizio Forte, PhD, Neuromed IRCCS
Other Study IDs: 6-2017
Record Dates: First submitted 2017-07-05; First posted 2017-07-07 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Aortic Aneurysm
Keywords: aortic aneurysm; autophagy; oxidative stress; Hippo pathway
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Aortic aneurysm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The molecular mechanisms contributing to the development of aortic aneurysmal disease are poorly characterized making actual therapies not sufficient. Autophagy is an intracellular mechanism that removes dysfunctional organelles and unfolded proteins, thereby maintaining cellular homeostasis. Activation of autophagy was shown to limit cardiac damage during stress. Accordingly, autophagy was found to be inhibited in the heart in animal models of metabolic syndrome, diabetes, obesity and aging thereby contributing to the development of cardiac derangements associated with these conditions. However, it remains to fully dissect the association between autophagy and structural alterations of the aortic wall and endothelial dysfunction in humans. In this study the correlation between levels of autophagy and the development of human aortic aneurysm will be assessed in patients subjected to surgical interventions for aortic pathologies. The association of Hippo signaling activation with the formation of aortic disease will also be evaluated, since previous work demonstrated that the Hippo pathway negatively regulates autophagy and promotes the development of cellular abnormalities. The results of this study may provide new insights into the mechanisms underlying the development of aortic disease.

DETAILED DESCRIPTION:
Autophagy may represent a new potential therapeutic target for the prevention and the treatment of aortic pathologies. It is a cellular self- digestion mechanism that prevents the accumulation of senescent organelles and damaged proteins. Autophagy plays a pivotal role in the regulation of cellular homeostasis and promotes the cellular response to stress. However, further investigations are needed to establish how autophagy is influenced by cardiovascular risk factors, as well as by pharmacological therapy. Moreover, it is still unclear in humans the association between autophagy and structural and functional alterations of aortic wall, as well as its association with endothelial dysfunction, especially in subjects affected by aortic pathologies. Furthermore, no data are available on the correlation between autophagy and the prognosis of patients who underwent cardio-surgical procedures for aortic pathologies. In this study, autophagy levels will be evaluated in human aortic aneurysm samples obtained from patients enrolled for a surgical aorta procedures. Autophagy markers in each aneurysm sample will be compared to those observed in the non-aneurysmatic aortic portion adjacent to the aneurysmatic tract obtained from the same patient. Levels of autophagy will also be correlated with markers of apoptosis and oxidative stress in both the aneurysmatic and non-aneurysmatic aortic parts. The involvement of the Hippo signaling pathway and inflammation in control and aneurysm samples will also be investigated. The investigators expect that autophagy levels will be lower in aneurysm samples with respect to non-aneurysmatic adjacent aortic portions. They will also be inversely correlated with aneurysm dimension. In contrast, the Hippo pathway will be activated in aortic aneurysms. Autophagy and Hippo signaling markers will also be correlated with markers of apoptosis and oxidative stress in aortic samples. In conclusion, the results of this study may underline the vascular role of autophagy and Hippo signaling and their involvement in the development of aortic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects undergoing aortic surgical procedures
* Ejection fraction (FE) > 30%
* Acceptance and signature of the informed consent

Exclusion Criteria:

* Acute myocardial infarction in the last 6 months
* Chronic and acute Inflammatory diseases
* Immunological and rheumatic diseases
* Pre-existing or ongoing neoplasms
* infectious diseases
* Treatment with pharmacological therapies able to modulate autophagy, i. e. rapamycin and derivative compounds (rapalogues))
* Antioxidant therapies in the last three months
* Patients with surgical technical complications

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects affected by abdominal aortic aneurysms undergoing aortic surgical procedures
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Comparison between the levels of Hippo signaling and autophagy markers observed in aortic aneurysms and the levels assessed in the adjacent non-aneurysmatic aortic portions. | 1 month
  Quantification by immunoblot of markers of Hippo signaling (MST1, YAP) and autophagy (LC3, p62, Beclin1, Atg5, Atg7, Ulk1. Adjacent aortic fragments without aneurysm belonging to the same patient will be used as control.

SECONDARY OUTCOMES:
Impact of cardiovascular risk factors on the autophagy levels in aortic samples of patients undergoing surgical procedure of aortic aneurysm removal. | 1 month
  Quantification by immunoblot of markers of autophagy (LC3, p62, Beclin1, Atg5, Atg7, Ulk1) and its statistical correlation with cardiovascular risk factors, such as age, diabetes, obesity, hypercholesterolemia, metabolic syndrome
Correlation between levels of autophagy and apoptosis in aneurysmal samples | 1 month
  Quantification by immunoblot of markers of autophagy and apoptosis
Correlation between levels of autophagy and endothelial function in patients undergoing surgical procedure of aortic aneurysm removal | 1 month
  flow- mediated dilatation (FMD) in subject underwent surgical procedure of aortic substitution/dissection
Correlation between levels of autophagy and the size of aortic aneurysms | 1 month
  Aneurysmal dimension will be evaluated by CT angiography

OTHER OUTCOMES:
Correlation between autophagy, oxidative stress and inflammation | 1 month
  western blot for markers of autophagy, ELISA and High Performance Liquid Chromatography (HPLC) analyses for markers of oxidative stress
Correlation between levels of autophagy and the Hippo pathway | 1 month
  western blot for marker of autophagy and the Hippo pathway

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Frati, MD, Principal Investigator — IRCCS Neuromed
Locations (1):
- IRCCS Neuromed, Pozzilli, Isernia, Italy